CLINICAL TRIAL: NCT04505878
Title: Vitamin C: Assessing Safety After Lung Transplant
Brief Title: Perioperative Vitamin C Lung Transplant
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Decided not to proceed with study
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0503; A530900 (Other: UW Madison); SMPH/ANESTHESIOLOGY (Other: UW Madison); Protocol Version 0.05 (Other: UW Madison)
Record Dates: First submitted 2020-08-05; First posted 2020-08-10 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Primary Graft Dysfunction; Lung Transplant; Complications
Keywords: Vitamin C
MeSH Terms: conditions — Primary Graft Dysfunction | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: This is a pilot single-arm unblinded trial to assess whether parenterally administered ascorbic acid (vitamin C) is safe in the lung transplant population.The investigators will not randomize or control; a retrospective cohort of participants not treated with vitamin C will be reviewed from 2015-2020. Those participants who decline the intervention will have the choice to consent to having their data be considered as part of the (non-retrospective) controls and be considered in our statistical analysis for outcomes, including analysis between this group and the historical controls. All participants who consent will be administered the therapy and participants will be evaluated via an intention-to-treat analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Vitamin C Arm (Experimental): Ascorbic Acid will be administered at a dose of 1500 mg in 100 mL of saline over 30 minutes intravenously once every 6 hours for a total of 72 hours
  Interventions: Drug: Vitamin C

INTERVENTIONS:
Drug: Vitamin C — Vitamin C is a first-line antioxidant that directly scavenges free radicals, inhibits reactive oxygen species (ROS) producing enzymes and recovers other cellular antioxidants
  Other Names: ascorbic acid

SUMMARY:
This study is being done to determine if parenterally administered ascorbic acid (Vitamin C) given at the time of lung transplant is safe. Vitamin C may be an effective intervention towards primary graft dysfunction (PGD). The study will enroll 69 participants who consent to the intervention. Participants who do not consent to the intervention will be treated according to standard-of-care, but may choose to be consented to have their data retrospectively reviewed. Based on our consent rate, this group may include 40-70 participants. Participants will be on study for up to 12 months.

DETAILED DESCRIPTION:
PGD is a frequent and severe outcome that impacts both short- and long-term outcomes after lung transplantation. Major pathophysiologic contributors include ischemia and reperfusion injury, mitochondrial dysfunction and endothelial failure. No directed therapy exists. Vitamin C is a first-line antioxidant that also acts at the endothelium and mitochondria to decrease permeability and leak, inhibit mitochondrial dysfunction and improve ischemia and reperfusion. When combined with steroids, part of standard care for lung transplant recipients, these effects may be enhanced and synergistically inhibit instigators of patient injury. A pilot trial will ensure safety of this potential intervention and guide future research into this important outcome measure. It will be readily received in the literature.

For the present study, vitamin C will be administered parenterally at a dose of 1,500 mg every 6 hours, a dose that is widely accepted and used in other clinical contexts where the drug is studied, such as sepsis. This will predictably reconstitute levels and achieve supratherapeutic benefit towards oxidant scavenging, while avoiding the potential pro-oxidant effects seen at exceedingly high doses. To this end, the investigators will exclude patients where the standard dosing of vitamin C will exceed 100 mg/kg/day (excluding patients <60 kg). Dosing will continue through post-operative day (POD) 3 to effectively assess for the impact of vitamin C on PGD.

Primary Objectives

* To assess whether parenterally administered ascorbic acid (vitamin C) is safe in the lung transplant population
* To estimate adherence to ascorbic acid administration protocol in this study population and to identify obstacles to feasibility of future trials using this protocol

Secondary Objectives

* To assess whether parenterally administered ascorbic acid (vitamin C) may decrease the rate and severity of PGD after lung transplant
* To establish the incidence of vitamin C and vitamin B1 (thiamine) deficiencies in the lung transplant population, and the responsiveness of vitamin C levels to our selected parenteral therapy
* To identify interventions that will optimize the post-operative wellbeing of patients receiving lung transplants by decreasing primary graft dysfunction (short and intermediate-to-long term

Stop Criteria

* Anuria x 3-hours
* Moderate, Grade 2 AKI (doubling of baseline creatinine)
* An acute, unexplained hemoglobin drop of >2 mg/dL

ELIGIBILITY:
Inclusion Criteria:

* Participant is scheduled for lung transplantation

Exclusion Criteria:

* Non-English speaking
* Subject is known or believed to be pregnant
* Subject is a prisoner.
* Subject has impaired decision-making capacity.
* Subject has known allergy to vitamin C.
* Subject has history of nephrolithiasis, oxalosis or hyperoxaluria. (Cystic Fibrosis patients are at risk of occult oxalosis / hyperoxaluria, therefore they will also be excluded from the study.)
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Sickle cell anemia
* Heredity hemochromatosis
* Baseline creatinine >2 mg/dL or any current kidney injury
* Weight <60 kg
* Vitamin C supplement use or administration (including HAT therapy) within the last month prior to transplantation
* Current enrolment in another research study
* Not suitable for study participation due to other reasons at the discretion of the investigators.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-04 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and Severity of Kidney Injury Post Operative Day (POD) 1 | Post Operative Day 1
  The primary endpoint is the safety of the vitamin C intervention. This will be measured by the incidence and severity of kidney injuries on POD 1, POD 2, POD 3, POD 4, and POD 7. Acute kidney injury (AKI) is defined as any creatinine (Cr) that is 1.5-times the participant's baseline / immediate preoperative creatinine. Severity escalates with increasing ratios: Mild, stage 1 AKI (Cr 1.5-1.99x baseline); Moderate, stage 2 AKI (Cr 2-2.9x baseline); and Severe, stage 3 AKI (Cr >3x baseline or any initiation of dialysis).
Incidence and Severity of Kidney Injury POD 2 | Post Operative Day 2
  The primary endpoint is the safety of the vitamin C intervention. This will be measured by the incidence and severity of kidney injuries on POD 1, POD 2, POD 3, POD 4, and POD 7. Acute kidney injury (AKI) is defined as any creatinine (Cr) that is 1.5-times the participant's baseline / immediate preoperative creatinine. Severity escalates with increasing ratios: Mild, stage 1 AKI (Cr 1.5-1.99x baseline); Moderate, stage 2 AKI (Cr 2-2.9x baseline); and Severe, stage 3 AKI (Cr >3x baseline or any initiation of dialysis).
Incidence and Severity of Kidney Injury POD 3 | Post Operative Day 3
  The primary endpoint is the safety of the vitamin C intervention. This will be measured by the incidence and severity of kidney injuries on POD 1, POD 2, POD 3, POD 4, and POD 7. Acute kidney injury (AKI) is defined as any creatinine (Cr) that is 1.5-times the participant's baseline / immediate preoperative creatinine. Severity escalates with increasing ratios: Mild, stage 1 AKI (Cr 1.5-1.99x baseline); Moderate, stage 2 AKI (Cr 2-2.9x baseline); and Severe, stage 3 AKI (Cr >3x baseline or any initiation of dialysis).
Incidence and Severity of Kidney Injury POD 4 | Post Operative Day 4
  The primary endpoint is the safety of the vitamin C intervention. This will be measured by the incidence and severity of kidney injuries on POD 1, POD 2, POD 3, POD 4, and POD 7. Acute kidney injury (AKI) is defined as any creatinine (Cr) that is 1.5-times the participant's baseline / immediate preoperative creatinine. Severity escalates with increasing ratios: Mild, stage 1 AKI (Cr 1.5-1.99x baseline); Moderate, stage 2 AKI (Cr 2-2.9x baseline); and Severe, stage 3 AKI (Cr >3x baseline or any initiation of dialysis).
Incidence and Severity of Kidney Injury POD 7 | Post Operative Day 7
  The primary endpoint is the safety of the vitamin C intervention. This will be measured by the incidence and severity of kidney injuries on POD 1, POD 2, POD 3, POD 4, and POD 7. Acute kidney injury (AKI) is defined as any creatinine (Cr) that is 1.5-times the participant's baseline / immediate preoperative creatinine. Severity escalates with increasing ratios: Mild, stage 1 AKI (Cr 1.5-1.99x baseline); Moderate, stage 2 AKI (Cr 2-2.9x baseline); and Severe, stage 3 AKI (Cr >3x baseline or any initiation of dialysis).
Incidence of New Dialysis Initiation | up to Post Operative Day 7

SECONDARY OUTCOMES:
Participant Vitamin C Levels | Baseline, Post Operative Day 1, Post Operative Day 2, Post Operative Day 3
Participant Thiamine Levels | Baseline, Post Operative Day 1, Post Operative Day 2, Post Operative Day 3
Incidence of Primary Graft Dysfunction (PGD) | up to Post Operative Day 7
  Primary Graft Dysfunction is defined as chest x-ray (CXR)-infiltrates with or without depressed oxygenation function, assessed by the "PF-Ratio," which is the PaO2 / FiO2.
Incidence and Severity of PGD on POD 3 | Post Operative Day 3
  Primary Graft Dysfunction is defined as chest x-ray (CXR)-infiltrates with or without depressed oxygenation function, assessed by the "PF-Ratio," which is the PaO2 / FiO2. Severity is defined as: PGD Grade 1 = CXR findings and any PF Ratio > 300; PGD Grade 2 = CXR findings and PF Ratio 200-300; and PGD Grade 3 = CXR findings and PF Ratio <200.
Tacrolimus Levels | Post Operative Days 2, 3, 4, and 7
Tacrolimus Doses | Post Operative Days 4 and 7
Post-Operative Well Being: Mortality | at Post Operative Day 30 and Post Operative Day 90 via chart review
Post-Operative Well Being: Atrial Fibrillation | up to Post Operative Day 7
Post-Operative Well Being: ICU Length of Stay | up to Post Operative Day 30 (chart review)
Post-Operative Well Being: Hospital Length of Stay | up to Post Operative Day 90 (chart review)
Post-Operative Well Being: Nadir Cardiac Index | up to 72 hours post op
Post-Operative Well Being: Peak Pulmonary Artery Systolic Pressure | up to 72 hours post op
Post-Operative Well Being: Peak Pulmonary Artery Diastolic Pressure | up to 72 hours post op
Post-Operative Well Being: Duration of Inotrope Need | up to 72 hours post op
Post-Operative Well Being: Duration of Vasopressor | up to 72 hours post op
Post-Operative Well Being: Total Dose of Vasopressor | up to 72 hours post op
Post-Operative Well Being: Daily Crystalloid Volume | up to 72 hours post op
  for 0-24h, 24-48h and 48-72h; total volume balance at 72-hours
Post-Operative Well Being: Daily Blood Product Transfusion Volume | up to 72 hours post op
  for 0-24h, 24-48h and 48-72h; total volume balance at 72-hours
Post-Operative Well Being: Daily Chest Tube Output Volume | up to 72 hours post op
  for 0-24h, 24-48h and 48-72h; total volume balance at 72-hours
Post-Operative Well Being: Duration of Post-Operative Mechanical Ventilation | up to Post Operative Day 7
Post-Operative Well Being: PaO2 / FIO2 ratios | Post Operative Day 1, Post Operative Day 2, Post Operative Day 3
  The PF Ratio assesses the lungs' ability to oxygenate the blood. It is defined as the ratio of the partial pressure of oxygen in the arteries (PaO2 in mmHg) to the fractional inspired oxygen content from the ventilator (FiO2 in %).
Post-Operative Well Being: Time to Clearance of Lactate | up to Post Operative Day 3
  "Clearance" is defined as a lactate <1 mmol/L.

CONTACTS AND LOCATIONS:
Overall Officials: Micah Long, MD, Principal Investigator — UW School of Medicine and Public Health

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be requested from other researchers up to 7 years after the completion of the primary endpoint by contacting Dr. Micah Long, the Principal Investigator of this study.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: up to 7 years after the completion of the primary endpoint